CLINICAL TRIAL: NCT06759909
Title: Influence of Use of Dapagliflozin on Outcomes of Rhythm Control Strategy (Pharmacological ± Interventional) in Patient with Atrial Fibrillation
Brief Title: Dapagliflozin on Outcomes of Rhythm Control Strategy (Pharmacological ± Interventional) in Patient with Atrial Fibrillation
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hanan Gamal, resident physician of cardiology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Dapagliflozin in AF Patients
Record Dates: First submitted 2024-12-22; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2025-01

CONDITIONS: Dapagliflozin (Forxiga); Atrial Fibrillation (AF)
Keywords: dapagliflozin; rythme control
MeSH Terms: conditions — Atrial Fibrillation | interventions — dapagliflozin

STUDY DESIGN:
Masking Description: We will record all baseline characteristics (Age, sex, BMI, HR and BP), AF type, EHRA class, previous use of ADD (B blockers, Class I, III AAD), previous CV, prior cerebrovascular stroke and Co-morbidities (HTN, DM, IHD, HF, Renal impairment, peripheral arterial disease, OSAS). CHADS2Vasc score and HAS-BLEED score will be calculated. Trans-thoracic echocardiograms will be performed within 4 weeks before the rhythm control attempts to determine LA diameter and volumes and left ventricular hypertrophy and functions (EF and E/'e).
  After enrollment, the patients will be treated with dapagliflozin (10 mg/d) or placebo at the time of rhythm control strategy and will continue daily treatment at the same dose till the 9 month follow-up period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dapagliflizon in Atrial fibrillation on Rythme control (Active Comparator): investigator study the efficacy and safety outcomes of Dapagliflozin use among newly diagnosed AF patients when underwent rhythm control strategy regardless their diabetic status.
  After enrollment, the patients will be treated with dapagliflozin (10 mg/d) or placebo at the time of rhythm control strategy and will continue daily treatment at the same dose till the 9 month follow-up period.
  Interventions: Drug: Dapagliflozin (DAPA)

INTERVENTIONS:
Drug: Dapagliflozin (DAPA) — We will record all baseline characteristics (Age, sex, BMI, HR and BP), AF type, EHRA class, previous use of ADD (B blockers, Class I, III AAD), previous CV, prior cerebrovascular stroke and Co-morbidities (HTN, DM, IHD, HF, Renal impairment, peripheral arterial disease, OSAS). CHADS2Vasc score and HAS-BLEED score will be calculated. Trans-thoracic echocardiograms will be performed within 4 weeks before the rhythm control attempts to determine LA diameter and volumes and left ventricular hypertrophy and functions (EF and E/'e).
  After enrollment, the patients will be treated with dapagliflozin (10 mg/d) or placebo at the time of rhythm control strategy and will continue daily treatment at the same dose till the 9 month follow-up period.

SUMMARY:
Investigator study the efficacy and safety outcomes of Dapagliflozin use among newly diagnosed Atrial fibrillation patients when underwent rhythm control strategy regardless their diabetic status.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common arrhythmia among adults with increasing risk of stroke, heart failure (HF) and mortality .

Based on the EAST-AFNET 4 trial and nationwide cohort studies, early rhythm control treatment (Antiarrhythmic drugs AAD or catheter ablation) was associated with a lower risk of adverse cardiovascular outcomes than usual care among patients who had recently (within one year) been diagnosed with atrial fibrillation A new oral hypoglycemic drug, dapagliflozin, a sodium-glucose cotransporter-2 inhibitor (SGLT2i), was confirmed to reduce the risk of cardiovascular adverse events (AEs) and improve coronary heart disease and HF outcomes in multiple clinical trials . In addition, previous post hoc analyses and meta-analyses reported that dapagliflozin can decrease the incidence rate of new-onset AF Recent trials and meta-analyses have reported that SGLT2i can achieve greater suppression of AF recurrence after catheter ablation (CA) in T2DM patients . Nonetheless, it remains unknown whether dapagliflozin can improve the recurrence of AF among newly diagnosed AF patients who underwent rhythm control strategy regardless the diabetic status.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed AF patients (Time between AF diagnosis to rhythm control attempt less than one year) Paroxysmal and persistent atrial fibrillation (AF) documented on a 12 lead ECG, Holter monitor (episodes of AF must be >30 seconds in duration to qualify as an inclusion criterion) Age of 18 years or older on the date of consent. Informed Consent

Exclusion Criteria:

* Long standing persistent AF. Previous use of dapagliflozin within one month of rhythm control attempt. Previous rhythm control attempt. AF due to reversible cause (e.g. hyperthyroidism, cardiothoracic surgery). History of congestive heart failure. Active intracardiac thrombus Pre-existing pulmonary vein stenosis or pulmonary vein stent Contraindication to anticoagulation or radio contrast materials

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-03 (Estimated); Primary Completion 2026-12-22 (Estimated); Study Completion 2028-12-22 (Estimated)

PRIMARY OUTCOMES:
freedom from any atrial arrhythmia | 9 month
  The primary effectiveness endpoint is freedom from any atrial arrhythmia (atrial arrhythmia defined as Atrial fibrillation or atrial tachycardia [AT] that lasted ≥ 30 seconds on/off AAD detected by the monitoring tools during the follow-up period excluding the first three months of the blanking period).

SECONDARY OUTCOMES:
cardiovascular hospitalization | 9 month
  Cardiovascular hospitalizations are defined as any hospitalizations due to cardiovascular cause such as AF related hospitalizations (such as emergency department (ED) visits, repeat ablation, electrical cardioversion and AV nodal ablation), device implantations, and decompensated HF hospitalization, stroke, myocardial infarction, vascular complications and major bleedings.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stachteas P, Karakasis P, Karagiannidis E, Patoulias D, Athanasiadou P, Nasoufidou A, Papadopoulos C, Kassimis G, Fragakis N. Efficacy of sodium-glucose cotransporter 2 inhibitors in preventing atrial fibrillation recurrence after catheter ablation. Hellenic J Cardiol. 2024 Sep-Oct;79:86-87. doi: 10.1016/j.hjc.2024.03.008. Epub 2024 Mar 12. No abstract available. PMID 38484841
- [Background] Luo F, Sun L, Wang Z, Zhang Y, Li J, Chen Y, Dong J. Effect of Dapagliflozin on the Outcome of Radiofrequency Catheter Ablation in Patients with Type 2 Diabetes Mellitus and Atrial Fibrillation. Cardiovasc Drugs Ther. 2024 Feb;38(1):91-98. doi: 10.1007/s10557-022-07368-2. Epub 2022 Aug 13. PMID 35962156
- [Background] Pluymaekers NAHA, Dudink EAMP, Luermans JGLM, Meeder JG, Lenderink T, Widdershoven J, Bucx JJJ, Rienstra M, Kamp O, Van Opstal JM, Alings M, Oomen A, Kirchhof CJ, Van Dijk VF, Ramanna H, Liem A, Dekker LR, Essers BAB, Tijssen JGP, Van Gelder IC, Crijns HJGM; RACE 7 ACWAS Investigators. Early or Delayed Cardioversion in Recent-Onset Atrial Fibrillation. N Engl J Med. 2019 Apr 18;380(16):1499-1508. doi: 10.1056/NEJMoa1900353. Epub 2019 Mar 18. PMID 30883054
- [Background] Packer DL, Mark DB, Robb RA, Monahan KH, Bahnson TD, Poole JE, Noseworthy PA, Rosenberg YD, Jeffries N, Mitchell LB, Flaker GC, Pokushalov E, Romanov A, Bunch TJ, Noelker G, Ardashev A, Revishvili A, Wilber DJ, Cappato R, Kuck KH, Hindricks G, Davies DW, Kowey PR, Naccarelli GV, Reiffel JA, Piccini JP, Silverstein AP, Al-Khalidi HR, Lee KL; CABANA Investigators. Effect of Catheter Ablation vs Antiarrhythmic Drug Therapy on Mortality, Stroke, Bleeding, and Cardiac Arrest Among Patients With Atrial Fibrillation: The CABANA Randomized Clinical Trial. JAMA. 2019 Apr 2;321(13):1261-1274. doi: 10.1001/jama.2019.0693. PMID 30874766